CLINICAL TRIAL: NCT05706311
Title: Adaption and Implementation of a Community Pharmacy-Based Prescription Drug Monitoring Program Opioid Risk Assessment Tool (PharmTool)
Brief Title: Community Pharmacy-Based Prescription Drug Monitoring Program Opioid Risk Assessment Tool
Acronym: PharmTool
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Cincinnati (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jerry Cochran, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTN-0138; 3UG1DA049444-04S2 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-01-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Opioid Abuse; Prescription Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a type-1 cluster 2-arm randomized trial. Randomization will take place at the pharmacy level and will be stratified by zip code level of poverty and pharmacy patient volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Pharmacy Site (Experimental): Pharmacies randomized to the experimental arm will be exposed to the intervention condition.
  Patients at the intervention pharmacy identified as at elevated risk will receive confirmatory screening for opioid risk. Those with confirmed moderate risk will receive a brief motivational intervention for medication misuse and an offer of naloxone dispensation. Those with high risk will receive a brief motivational intervention leading to warm handoff treatment linkage intervention to primary or specialty substance use care with an offer for naloxone dispensation.
  Interventions: Behavioral: Clinical Decision Support Tool (Moderate Risk); Behavioral: Clinical Decision Support Tool (High Risk)
- Control Pharmacy Site (Other): Standard of Care is the treatment as usual condition, which follows federal and Ohio state pharmacy requirements for pharmacists where in patients filling prescriptions receive information and opt-in counseling. Ohio State law requires pharmacist to not dispense an opioid supply >90 days, with a specific prohibition on dispensations ≥14 days after prescriptions are issued. Pharmacists are also required to perform a universal prescription drug medication review before initial dispensation and offer brief counseling (e.g., unstandardized information about medication safety) for new/modified prescription therapies.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Clinical Decision Support Tool (Moderate Risk) — Moderate risk patients will get brief motivational intervention for medication misuse and an offer of naloxone dispensation.
  Arms: Intervention Pharmacy Site
Behavioral: Clinical Decision Support Tool (High Risk) — Those with high risk will receive a brief motivational intervention leading to warm handoff treatment linkage intervention to primary or specialty substance use care with an offer for naloxone dispensation.
  Arms: Intervention Pharmacy Site
Other: Standard of Care — Ohio State law requires pharmacist to not dispense an opioid supply >90 days, with a specific prohibition on dispensations ≥14 days after prescriptions are issued. Pharmacists are also required to perform a universal prescription drug medication review before initial dispensation and offer brief counseling (e.g., unstandardized information about medication safety) for new/modified prescription therapies.
  Arms: Control Pharmacy Site

SUMMARY:
This goal of this observational study is to develop and test the Opioid Risk Reduction Clinical Decision Support (ORRCDS) tool. The tool will be an opioid medication risk screener and decision support platform that will be used by pharmacists upon dispensing prescription opioid medication. Once the Opioid Risk Reduction has been developed, we will examine the impact of the ORRCDS within two divisions of a large chain retail pharmacy. Pharmacies will be randomized to using the Opioid Risk Reduction Clinical Decision Support (ORRCDS) tool or standard of care opioid dispensation. We hypothesize that patients at pharmacies randomized to the ORRCDS tool will be more likely to reduce their risk status to low or moderate compared to the patients at standard of care pharmacies.

DETAILED DESCRIPTION:
In our previous research, patients have reported a willingness to answer questions and discuss opioid medication use with pharmacists in these settings. Therefore, community pharmacy settings are an underused resource with great promise for screening and engaging patients to reduce opioid medication misuse. Currently, prescription drug monitoring programs (PDMP) are the most available tool to pharmacists for monitoring opioid use among patients. As a result, PDMP users must rely on their "best judgment" in clinical decision-making and often provide patient care and referrals with a limited evidence base. The question of highest importance in the field of prescription medication misuse is: How can PDMP information/output be most usefully utilized for patient intervention within an evidence-based opioid risk reduction clinical decision support (ORRCDS) tool.

This study will develop and test the Opioid Risk Reduction Clinical Decision Support (ORRCDS) tool and examining facilitators and barriers to sustainability and broader dissemination. The study is organized into 3 aims:

Aim 1: ORRCDS Tool development which will include a universal opioid medication risk screener and decision support platform.

Aim 2: Once the ORRCDS has been developed, we will conduct a type-1 cluster 2-arm randomized trial to examine the impact of the ORRCDS tool within two divisions of a large chain retail pharmacy. We hypothesize that patients with moderate or high opioid risk will be more likely to reduce risk status to low or moderate following ORRCDS implementation compared to standard care.

Aim 3: Following the completion of the cluster randomized trial, qualitative interviews will be conducted with pharmacists and leaders from a large chain retail pharmacy and PDMP vendor about the potential barriers and facilitators to the sustainability (continued use at the stores in this project) and broader dissemination (implementation at other stores outside of those in this project) of the ORRCDS.

ELIGIBILITY:
Inclusion Criteria:

* A large chain retail pharmacy chain in the Cincinnati or Columbus, Ohio area

Exclusion Criteria:

* None

This study does not involve individual patients as randomization will occur among pharmacies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Development of the Opioid Risk Reduction Clinical Decision Support (ORRCDS) tool | 24 months
  This outcome will be assessed using the System Usability Scale (SUS).
Stage 2: Improvement in patient opioid-related risks | 24 months
  This outcome will be assessed using the Narcotic Score (NS).
Stage 3: ORRCDS sustainability within the system and pharmacy chain systems | 24 months
  Using the Consolidated Framework for Implementation Research the investigators will interview staff from the PDMP vendor and large chain retail pharmacy to assesses the barriers of tool sustainability.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cochran, PhD, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No